CLINICAL TRIAL: NCT06436989
Title: Effect of Temperature Leaching Solution of Disposable Plastic Tableware on Intestinal Health of Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang Zeng (Other Government)
Responsible Party: Sponsor-Investigator, Xiang Zeng, Associate professor, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 20240306-1
Record Dates: First submitted 2024-05-06; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Intestinal Dysfunction; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hot water (Experimental): 300ml pure water cooled to room temperature in a kettle.
  Interventions: Other: hot purified water
- normal temperature water (Placebo Comparator): 300 ml pure water without any treatment
  Interventions: Other: hot purified water

INTERVENTIONS:
Other: hot purified water — Hot purified water,drink once a workday,almost 360mL.Buy from regular channels.

SUMMARY:
Studies have shown that disposable plastic tableware will cause harm to human health after heat exposure, which is closely related to the rapid development of modern society and economy and the accelerated pace of life. Most of the existing studies focused on the characterization of micro-nano plastic particles and organic pollutants such as bisphenol A and polycyclic aromatic hydrocarbons produced after thermal exposure of disposable plastic tableware, but did not pay sufficient attention to the potential relationship with individual health effects. In addition; Sporadic animal tests and molecular tests have verified the health hazards of disposable plastic tableware leaching solution. Based on the previous research results, we believe that the leaching solution of disposable plastic tableware at high temperature environment will disturb the intestinal flora structure, affect the intestinal metabolic profile, and produce adverse health outcomes for human intestinal health. This study intends to recruit healthy school students as research objects, and collect urine and stool samples of test subjects, in order to explore the effects of high-temperature leaching solution of disposable plastic tableware on intestinal health of adults.

DETAILED DESCRIPTION:
The method of single blind randomized controlled cross trial was adopted. A total of 80 healthy adults were recruited and divided into test group and control group according to the principle of randomization. During the trial period, the experimental group used a disposable plastic cup to drink a cup of hot water boiled in a hot kettle in the morning and in the evening (reduced to room temperature, about 300mL), while the control group also used a disposable plastic cup to drink room temperature water without heat exposure. The first phase lasted for 5 working weeks, and after a one-month washout period in the middle, the experimental group and the control group crossed. The second phase of the cross-over trial also lasted 5 workweeks. A total of four medical examinations were performed throughout the trial period, before and after the first and second trials. A check-up lasts half a day.

Health outcome indicators: height, weight, body composition analysis, saliva, blood pressure, blood, urine sample, stool sample indicators.

Urine, feces and blood samples were collected to detect the relevant indicators in order to explore the potential mechanism of the harm of heavy metals in the hot exposure leaching solution of disposable plastic tableware to human intestinal health.

ELIGIBILITY:
Inclusion Criteria:

* .Healthy college students aged 18 to 35;
* .Subjects can receive the intervention in this study.

Exclusion Criteria:

* 1.Have been diagnosed with diabetes, ulcerative colitis, Crohn's disease, or an infectious disease;

  * Chemotherapy, radiation or surgery 3-6 months prior to sampling;
  * Abnormal bowel movements one week before sampling;
  * I was menstruating at the time of sampling;
  * In the past three months, the sample has taken probiotics and other related health products and dietary supplements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity(FVC) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4weeks plants exposure in second stage
  We plan to measure forced vital capacity (FVC) of lung function.
Blood Pressure(BP) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4weeks plants exposure in second stage.
  We plan to measure systolic blood pressure (SBP) and diastolic blood pressure (DBP)

SECONDARY OUTCOMES:
Heart Rate Variability(HRV) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4weeks plants exposure in second stage.
  We plan to measure Heart Rate Variability (HRV).

OTHER OUTCOMES:
C-reactive protein(CRP) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4weeks plants exposure in second stage.
  We plan to measure serum concentrations of C-reactive protein(CRP)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Chinese Medicine University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided